CLINICAL TRIAL: NCT02108821
Title: A Study of Fecal Microbiota Transplantation in Pediatric Patients With Relapsed Inflammatory Bowel Disease.
Brief Title: Fecal Microbiota Transplantation in Pediatric Patients
Acronym: FMT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Pittsburgh (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO13030081
Record Dates: First submitted 2014-03-21; First posted 2014-04-09 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Inflammatory Bowel Diseases (IBD); Crohn's Disease (CD); Ulcerative Colitis (UC)
Keywords: Inflammatory Bowel Diseases (IBD); Crohn's Disease (CD); Ulcerative Colitis (UC)
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal Microbiome Transplantation (Experimental): Fecal Microbiome Transplantation will be done at the time of EGD and colonoscopy. A parent or sibling or a healthy relative will be tested for several infections like hepatitis, H. Pylori, HIV, syphilis, ova and parasites, culture and C.diff. They will fill out a donor questionnaire used for blood donors prior to the sample collection. After eligibility criteria have been met, appropriate consent has been obtained, and the screening labs have been assessed, the fecal transplant procedure will take place in the procedure center at Children's Hospital of Pittsburgh. Fresh stool sample will be obtained from the donor. The fecal sample will be prepared for transplantation in a designated area in the procedure center. Frequency: once. Duration: Approximately 1 hour
  Interventions: Biological: Fecal Microbiota Transplantation (FMT)

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation (FMT) — The process of fecal microbiota transplantation (FMT), where fecal bacteria from a healthy individual is transferred into a recipient as an alternative therapy for individuals affected with these life-altering diseases: Crohn's Disease (CD), and/or Ulcerative Colitis (UC).
  Other Names: Fecal Transplantation

SUMMARY:
A disturbance in the diversity of gut bacterial composition could be linked to several immune mediated diseases including inflammatory bowel diseases (IBD). IBD can be classified into Crohn's Disease (CD) and Ulcerative Colitis (UC). Both these diseases occur from abnormal immune reaction to resident gut bacteria.The process of fecal microbiota transplantation (FMT) where fecal bacteria from a healthy individual is transferred into a recipient, has recently received attention as an alternative therapy for individuals affected with these life-altering diseases. In this study, the investigators will perform fecal transplantation on the subjects meeting inclusion criteria, to determine the efficacy and safety of this therapy in subjects with IBD (CD and UC) who are not responding to first line therapy, and are in a flare.

DETAILED DESCRIPTION:
50 subjects (25 subjects with Crohn's Disease and 25 subjects with Ulcerative Colitis) who are 2 to 22 years of age will be enrolled in the trial over 3 years. The fecal donors, preferably a parent or sibling, will be extensively screened for infectious diseases prior to providing stool for the transplant. Patients who are failing primary therapy, are in a flare, and require restaging of their IBD by an endoscopy and colonoscopy will be approached for the study. Standard of care endoscopy and colonoscopy will be performed on each subject and 2 additional biopsies will be taken for analysis. Microbiota analysis will also be performed on both the donor and recipient stool sample prior to transplantation, and on the recipient sample at 1 week, 1 month, and 6 months post transplantation. The primary objective will be to study the safety of FMT in all enrolled subjects. The study will also correlate efficacy and patient outcomes with the fecal microbiome prior to, and after FMT. The secondary objectives are to examine the efficacy of FMT in the treatment of children with IBD using the Pediatric Ulcerative Colitis Activity Index (PUCAI) and the Pediatric Crohn Disease Activity Index (PCDAI) analysis. Correlate the patient outcomes with the fecal microbiome prior to, and after FMT.

ELIGIBILITY:
STUDY SUBJECT INCLUSION CRITERIA:

Current IBD patients who have:

* UC patients with a flare due to failure of current therapy and have to undergo esophagogastroduodenoscopy (EGD) and colonoscopy for restaging the disease and escalation of therapy.
* CD patients with ileo colonic or colonic disease who require an EGD and colonoscopy for disease assessment due to a flare or poor control.
* The ability to safely undergo colonoscopy (physical status classification used by the American Society of Anesthesiologists).
* PUCAI score less than sixty five.
* PCDAI score less than forty.

STUDY SUBJECTS EXCLUSION CRITERIA:

* Patients with Crohn's disease: complications like an abscess, phlegmon, stricture, small bowel obstruction, perforation, internal or external fistulization or infection as causes for flare up before being deemed eligible for recruitment to the study. We will check for these complications if a recent study has not been done.
* Severe immunosuppression: Biologicals with concomitant steroids (>30 mg/day).
* Central Line.
* Pressor or ventilatory support.
* On antibiotics.
* Patients with Crohn's disease found to have complications like an abscess, phlegmon, stricture, small bowel obstruction, perforation, internal or external fistulization or infection.
* Not willing to consent or follow guidelines throughout research trial.
* Screening labs in either donor or recipient reveal problems with performing fecal microbiome transplantation because inclusion requirements are no longer met.
* Physician discretion.
* Participant request.

DONOR EXCLUSION CRITERIA:

* A history of antibiotic treatment during the 3 months preceding donation.
* A history of intrinsic gastrointestinal illnesses.
* A history of autoimmune or atopic illness or modulating therapy.
* A history of chronic pain syndromes, or neurologic or neurodevelopmental disorders.
* Metabolic syndrome or malnutrition or obesity.
* A history of exposure to infectious agents.
* Diarrhea or other symptoms of an intestinal infection within two weeks prior to, or on the day of, stool donation.
* A history of malignant illnesses or ongoing oncologic therapy.
* Weight less than 15 kgs.

Ages: 2 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alka Goyal, MD, Principal Investigator — Stanford University
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fecal Microbiome Transplantation-open Label: Fecal Microbiome Transplantation will be done at the time of EGD and colonoscopy. A parent or sibling or a healthy relative will be tested for several infections like hepatitis, H. Pylori, HIV, syphilis, ova and parasites, culture and C.diff. They will fill out a donor questionnaire used for blood donors prior to the sample collection. After eligibility criteria have been met, appropriate consent has been obtained, and the screening labs have been assessed, the fecal transplant procedure will take place in the procedure center at Children's Hospital of Pittsburgh. Fresh stool sample will be obtained from the donor. The fecal sample will be prepared for transplantation in a designated area in the procedure center. Frequency: once. Duration: Approximately 1 hour
  Fecal Microbiota Transplantation (FMT): The process of fecal microbiota transplantation (FMT), where fecal bacteria from a healthy individual is transferred into a recipient as an alternative therapy for individuals affected
Period: Overall Study
Arm/Group | Fecal Microbiome Transplantation-open Label
Started (March 12, 2014) | 23
Completed (September 30th, 2016) | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Fecal Microbiome Transplantation: Use of Fecal Microbiome Transplantation for participants with IBD.
Arm/Group | Fecal Microbiome Transplantation
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 10 [8 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Outpatient Gastroenterology clinic Children's Hospital of Pittsburgh. Pittsburgh. Pennsylvania. USA
  Participants
    United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Occurrences of Adverse Events at 6 Months According to Adverse Event Term
Description: Adverse events recorded to determine safety of Fecal Microbiome Transplant in the treatment of children with IBD.
Time Frame: 6 months
Measure: Number; unit: Events
Groups:
- Overall Study: Overall Study Events
Arm/Group | Overall Study
Number analyzed (Participants) | 21
Events
  Moderate Abdominal Pain | 11
  Diarrhea | 5
  Flatulence and Bloating | 5
  Emesis | 3
  Bloody Stools | 2
  Nausea | 2
  Fever | 1

2. Secondary Outcome: Examine the Efficacy of Fecal Microbiome Transplant in the Treatment of Children With IBD Using the Pediatric Ulcerative Colitis Activity Index (PUCAI) and the Pediatric Crohn Disease Activity Index (PCDAI) Analysis.
Description: Efficacy outcomes scored via Pediatric Ulcerative Colitis Activity Index (PUCAI) and the Pediatric Crohn Disease Activity Index (PCDAI) analysis.
  Scored at baseline, day 30, and at day 180 for responders.
  The PUCAI score range is 0-85, where the higher the number the more severe the disease (A score of 65 and up is considered severe, a score of 35-64 is considered moderate, and a score of 10-34 is considered mild). The PUCAI is the scoring system used for patients with ulcerative colitis/indeterminate colitis.
  The PCDAI score range is 0-100, where the higher the number the more severe the disease (A score of greater than 30 is considered moderate to severe, a score of 11-30 is considered mild, and a score of 10 or less is considered inactive disease). The PCDAI is the scoring system used for patients with crohn's disease.
Time Frame: Baseline, Day 30, Day 180
Population: Only participants that responded to treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Fecal Microbiome Transplantation Ulcerative Colitis/Indeterminate Colitis: Use of Fecal Microbiome Transplantation for participants with Ulcerative Colitis/Indeterminate Colitis.
- Fecal Microbiome Transplantation With Crohn's Disease: Use of Fecal Microbiome Transplantation for participants with Crohn's Disease.
Arm/Group | Fecal Microbiome Transplantation Ulcerative Colitis/Indeterminate Colitis | Fecal Microbiome Transplantation With Crohn's Disease
Number analyzed (Participants) | 3 | 3
score on a scale
  Baseline | 40 [38.04 to 41.96] | 11.6 [9.64 to 13.56]
  Day 30 in responders | 11.6 [9.64 to 13.56] | 1.6 [0 to 3.56]
  Day 180 in responders | 21.6 [19.64 to 23.56] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Fecal Microbiota Transplantation: Use of Fecal Microbiota Transplantation for participants with IBD.
Arm/Group | Fecal Microbiota Transplantation
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 12/23
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fecal Microbiota Transplantation (N=23)
Abdominal Pain (Gastrointestinal disorders) | 11
Diarrhea (Gastrointestinal disorders) | 5
Flatulence and bloating (Gastrointestinal disorders) | 5
Emesis (Gastrointestinal disorders) | 3
Bloody stools (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Fever (General disorders) | 1

LIMITATIONS AND CAVEATS:
small number of subjects, open label trial, fecal calprotectin not collected in every subject so response measurement was subjective

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT02108821/Prot_SAP_000.pdf